CLINICAL TRIAL: NCT02244346
Title: Secotex®: Prescription Event Monitoring in Patients With Benign Prostatic Hyperplasia (BPH)
Brief Title: Prescription Event Monitoring in Patients With Benign Prostatic Hyperplasia (BPH)
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 527.58
Record Dates: First submitted 2014-09-18; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Benign prostatic hyperplasia patients
  Interventions: Drug: Secotex®

INTERVENTIONS:
Drug: Secotex®

SUMMARY:
Study to evaluate the safety profile of Secotex® in the improvement of the symptoms of Benign Prostatic Hyperplasia in real clinical practice

ELIGIBILITY:
Inclusion Criteria:

* Patients of any age with a diagnosis of symptomatic Benign Prostatic Hyperplasia (BPH)
* Patients with symptoms, that according to physician require medical treatment to improve quality of life
* Patients could be naive to treatment or could be on treatment with other drugs but have not responded adequately to treatment

Exclusion Criteria:

* Patients with known hypersensitivity to Tamsulosin, or any other component of the product
* Patients with a history of orthostatic hypotension or severe liver failure

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with Secotex® in the daily clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 811 (Actual)
Dates: Start 2004-05; Primary Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | up to 6 months